CLINICAL TRIAL: NCT07310706
Title: Eight-Week, Single-Site Study to Evaluate the Efficacy of a Facial Sunscreen in Adult Participants With Oily Skin and Signs of Aging
Brief Title: A Study to Evaluate the Efficacy of a Facial Sunscreen in Adult Participants With Oily Skin and Signs of Aging
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kenvue Brands LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CS2025SK100253
Record Dates: First submitted 2025-11-20; First posted 2025-12-30 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12-18

CONDITIONS: Oily Skin Aging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I: 30 to 44 years of age (Experimental): Group I: 30 participants in the age group of 30 to 44 years old, being:
  * At least 8 with skin type I and II on the Fitzpatrick scale
  * At least 8 with skin type III and IV on the Fitzpatrick scale
  * At least 8 with skin type V and VI on the Fitzpatrick scale
  Interventions: Other: Sunscreen A use
- Group II: 45 to 55 years of age (Experimental): Group II: 30 participants in the age group of 45 to 55 years old, being:
  * At least 8 with skin type I and II on the Fitzpatrick scale
  * At least 8 with skin type III and IV on the Fitzpatrick scale
  * At least 8 with skin type V and VI on the Fitzpatrick scale
  Interventions: Other: Sunscreen A use

INTERVENTIONS:
Other: Sunscreen A use — The application of the Investigational Product will be performed by the participant and supervised by a qualified technician at Visit 1 and by the participant in their home.
  Home use:
  The Investigational Product will be applied topically by the participant, following the following mode of use:
  "Apply an abundant amount (equivalent to one teaspoon) daily to the face and neck, at least twice a day, with reapplications whenever necessary."

SUMMARY:
This is a Single-Site, open-label, randomized clinical study that aims to evaluate the efficacy of the investigational product in improving the signs of skin aging and reducing facial oiliness in a population from 30 to 55 years of age.

ELIGIBILITY:
Inclusion Criteria:

1. For group I: 30 to 44 years of age; For group II: 45 to 55 years of age;
2. Skin Type I to VI according to Fitzpatrick's classification. For each group:

   I. Fitzpatrick I and II: at least 8 participants II. Fitzpatrick III and IV: at least 8 participants III. Fitzpatrick V and VI: at least 8 participants
3. Participants of any ethnicity according to IBGE criteria;
4. Participants with oily or combination skin and oily shine on the face, both self-declared (through applied questionnaire) and confirmed by the dermatologist (from 2 points for oil shine by the modified Griffith scale from 0 to 9) at inclusion. For group I: oiliness will also be confirmed by Sebumeter (value above 100 AU for inclusion);
5. Participants self-declared to have enlarged pores, confirmed by dermatologist;
6. Participants who show signs of mild to moderate aging (2 to 6 points for the parameters of wrinkles, fine lines, and skin roughness based on the modified Griffith scale of 0-9 points), confirmed by dermatologist at inclusion;
7. Participant reports, at the time of inclusion, that he/she is concerned with at least one of the following parameters related to the appearance of facial skin:

   I. Fine lines II. Wrinkles III. Roughness/uneven texture
8. Good general health, based on participant-reported medical history;
9. Able to read, write, speak and understand Portuguese;
10. For male participants: agree to shave 48 hours before study visits;
11. Person who signed the ICF and ICIU;
12. Intend to complete the study and are willing and able to follow all the instructions of the study.

Exclusion Criteria:

1. Have known allergies or adverse reactions to common topical skin care products, including facial sunscreen;
2. Have a skin condition that may influence the outcome of the study (specifically psoriasis, eczema, atopic dermatitis, cutaneous xerosis, erythema, or active skin cancer);
3. Present primary/secondary lesions (e.g., scars, ulcers, vesicles, irritation resulting from the removal of facial hair) in the test areas;
4. Report having Type 1 or Type 2 diabetes or taking insulin or other antidiabetic medication;
5. Using medications that could mask an adverse event (AE) or influence the results of the study, including:

   * Immunosuppressive or steroidal medications within 2 months prior to the first visit
   * Non-steroidal anti-inflammatory drugs within 5 days prior to the first visit
   * Antihistamines within 2 weeks prior to the first visit
   * Antibiotics (oral or topical), hormonal therapy (except hormonal contraception methods), insulin, inhaled steroids (except prescribed for temporary allergy relief) within 1 month prior to the first visit.
6. Participants who have undergone invasive aesthetic or dermatological treatments in the test area (face) within 2 months prior to the first visit;
7. Menopausal or postmenopausal women (except for perimenopausal women who are eligible for the study);
8. Presence of excess hair in the evaluation area (face) that may interfere with instrumental evaluations. In the case of men, they will be instructed to shave 48 hours before visits;
9. Use of any products that may interfere with study assessments, at the discretion of the dermatologist;
10. Participants who have undergone chemical and/or physical peeling, laser, or similar aesthetic treatments within 6 months prior to the study;
11. Participants who reported being pregnant, planning to become pregnant, or breastfeeding during the study;
12. Have a history of or currently have a health condition/situation that could put the subject at significant risk, confound the results of the study, or significantly interfere with their participation in the study;
13. Be simultaneously participating in another clinical study;
14. Be an employee/contractor or close relative of the PI, Study Site or Sponsor;
15. Participants who practice activities (leisure or work) with intense sun exposure;
16. Smoking participants (Note: participants living with smokers may be eligible, provided that, at the discretion of the investigator, the participant's exposure to cigarettes does not interfere with or confound the results of the study. The participant's coexistence with a smoker must be reported as informative data).

Ages: 30 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 73 (Actual)
Dates: Start 2025-08-21 (Actual); Primary Completion 2025-10-16 (Actual); Study Completion 2025-11-26 (Actual)

PRIMARY OUTCOMES:
Clinical efficacy of the use of Investigational Product on signs of facial aging via dermatological evaluation | Before and after Visit 1 (Day 0), Visit 2 (28 ± 2 days) and Visit 3 (56 ± 2 days ) of IP use
  It is expected to obtain statistical improvement (p≤0.05) in the evaluated attributes such as reduction of wrinkles, fine lines and roughness of the skin through the dermatological clinical evaluation of wrinkles, fine lines, and skin roughness parameters using the modified 10-point Griffith scale (from 0 to 9).
Clinical efficacy of Investigational Product in reducing skin oiliness via dermatological evaluation | Before and after Visit 1 (Day 0), Visit 2 (28 ± 2 days) and Visit 3 (56 ± 2 days ) of IP use
  It is expected to obtain statistical improvement (p≤0.05) in the evaluated attributes such as reduction of oiliness, reduction of oiliness shine, reduction of the appearance of pores through the dermatological clinical efficacy of oil shine using the modified 10-point Griffith scale (from 0 to 9).
Clinical efficacy of Investigational Product in reducing pores | Before and after Visit 1 (Day 0) and Visit 3 (56 ± 2 days ) of IP use
  It is expected to obtain statistical improvement (p≤0.05) in the evaluated attributes such as reduction of the appearance of pores through the dermatological clinical efficacy of pore appearance via modified 10-point Griffith scale (from 0 to 9).
Efficacy perceived by the participant through a questionnaire assessment | Before and after Visit 1 (Day 0) and Visit 3 (56 ± 2 days ) of IP use
  Efficacy measured by the participant through a questionnaire evaluating:
  * clinical efficacy of the use of Investigational Product on signs of facial aging
  * clinical efficacy of Investigational Product in reducing skin oiliness
  * clinical efficacy of Investigational Product in reducing pores
Clinical efficacy of the use of Investigational Product on signs of facial aging | Before and after Visit 1 (Day 0) and Visit 3 (56 ± 2 days ) of IP use
  Facial image captures using the COLORFACE equipment.
Clinical efficacy of the use of Investigational Product on signs of facial aging via image analysis | Before and after Visit 1 (Day 0), Visit 2 (28 ± 2 days) and Visit 3 (56 ± 2 days ) of IP use
  It is expected to obtain statistical improvement (p≤0.05) in the evaluated equipment described below:
  - Evaluation of the facial images by the ANTERA 3D equipment.
Clinical efficacy of Investigational Product in reducing skin oiliness via instrumental measurements | Before and after Visit 1 (Day 0), Visit 2 (28 ± 2 days) and Visit 3 (56 ± 2 days ) of IP use
  It is expected to obtain statistical improvement (p≤0.05) in the evaluated attributes such as reduction of oiliness through the equipment below:
  * Instrumental measurements with the Sebumeter® equipment.

SECONDARY OUTCOMES:
The clinical efficacy of Investigational Product in maintaining skin hydration | Before and after Visit 1 (Day 0) and Visit 3 (56 ± 2 days ) of IP use
  It is expected to obtain statistical improvement (p≤0.05) in the evaluated attributes, such as skin hydration through the equipment and evaluations described below:
  - To evaluate the clinical efficacy of Investigational Product in maintaining skin hydration, by measurements with Corneometer® equipment.
The clinical efficacy of Investigational Product in maintaining the skin barrier | Before and after Visit 1 (Day 0) and Visit 3 (56 ± 2 days ) of IP use
  It is expected to obtain statistical improvement (p≤0.05) in the evaluated attributes, such as reduction and/or maintenance of trans epidermal water loss through the equipment and evaluations described below:
  - To evaluate the clinical efficacy of Investigational Product in maintaining trans epidermal water loss with Tewameter equipment.

CONTACTS AND LOCATIONS:
Locations (1):
- CIDP do Brasil Pesquisas Clínicas LTDA, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: No